CLINICAL TRIAL: NCT04548648
Title: LCCC1841: A Pilot Study of Acalabrutinib in Relapsed/Refractory Primary and Secondary CNS Lymphomas
Brief Title: A Pilot Study of Acalabrutinib in Relapsed/Refractory Primary and Secondary CNS Lymphomas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1841
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Central Nervous System Lymphoma
Keywords: CNS Lymphoma
MeSH Terms: interventions — acalabrutinib

STUDY DESIGN:
Intervention Model Description: Simon Two-stage study to a pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label, single-arm (Other): A multicenter open-label, single-arm, phase 2 study designed to investigate the antitumor effects of acalabrutinib in subjects with relapsed primary central nervous system lymphoma (PCNSL), and relapsed secondary CNS lymphoma (SCNSL) with no evidence of current systemic disease. Subjects will receive acalabrutinib at the dose of 100 mg every 12 hours.
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib at 100 mg is taken orally approximately every 12 hours until disease progression or unacceptable toxicity.
  Other Names: ACP-196; CALQUENCE

SUMMARY:
The purpose of this study is to test whether giving acalabrutinib is safe and effective in controlling relapsed central nervous system (CNS) lymphoma. Currently, there are no FDA-approved treatments for relapsed CNS lymphoma. Although acalabrutinib has not been approved for the treatment of CNS lymphoma, it was approved for the treatment of another type of lymphoma (mantle cell), by the Food and Drug Administration (FDA).

Acalabrutinib acts similar to another cancer drug called ibrutinib. lbrutinib was tested in several research trials for the management of CNS lymphomas, and the results were promising. Acalabrutinib and ibrutinib attack a similar target found in CNS lymphoma. Acalabrutinib may do a better job in attacking this target than ibrutinib. The study doctors will be looking to see if acalabrutinib can shrink cancer cells.

DETAILED DESCRIPTION:
This multicenter open-label, single-arm, pilot study explores a safe and effective treatment for relapsed central nervous system lymphoma. The study investigates the antitumor effects and safety of acalabrutinib in subjects with relapsed primary central nervous system lymphoma (PCNSL) or relapsed secondary CNS lymphoma (SCNSL) with no evidence of current systemic disease. Types of SCNSL included in the study are: Diffuse large B-cell lymphoma, mantle cell lymphoma, plasmablastic lymphoma, and lymphoplasmacytic lymphoma. Up to 16 subjects will be enrolled to attain a total of 15 evaluable subjects.

Duration of Follow-up All subjects will be followed for survival for 5 years or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to participate in all required evaluations and procedures in this study protocol, including swallowing capsules and tablets without difficulty.
2. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).
3. Age ≥18 years at the time of consent.
4. Subject has adequate performance status as defined by The Eastern Cooperative Oncology Group (ECOG) of ≤ 2
5. Subject has histological confirmation of biopsy-proven central nervous system (CNS) lymphoma or magnetic resonance imaging (MRI) findings consistent with CNS lymphoma if biopsy is not possible (due to inaccessible location). Subjects with intra-ocular lymphoma will not be excluded as long as there is also parenchymal disease.
6. Subject has B-cell Non-Hodgkin Lymphoma.
7. Subject has no evidence of systemic involvement of lymphoma confirmed by computerized tomography (CT) or positron emission tomography (PET)-CT imaging within 28 days prior to first dosing in the study.
8. Subject must have received at least one prior line of chemotherapy for primary or secondary CNS lymphoma.
9. Subject has adequate organ function as demonstrated by: System Laboratory Value Hematological* Absolute Neutrophil Count (ANC) ≥ 1 x 109/L Platelets ≥ 75 x 109/L Renal* Calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault formula (Appendix B) Hepatic* Bilirubin ≤ 1.5 × upper limit of normal (ULN). Subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level >1.5 mg/dL if their conjugated bilirubin is <1.5× ULN) Aspartate aminotransferase (AST) ≤ 2.5 × ULN Alanine aminotransferase (ALT) ≤ 2.5 × ULN Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) and Activated Partial Thromboplastin Time (aPTT) ≤ 2 × ULN (in the absence of lupus anticoagulant)

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will not be able to participate in this study.

1. Prior cancer treatment that was completed less than 14 days prior to Day 1 of study dosing or if subject has not recovered from all reversible acute toxic effects of the regimen to grade ≤1 or baseline.
2. Prior brain radiotherapy under the following conditions:

   * Whole-brain radiotherapy (WBRT) that was completed less than 28 days prior to Day 1 of study dosing
   * Stereotactic radiosurgery (SRS) that was competed less than 14 days prior to Day 1 of study dosing.
3. Currently participating in or has participated in a study of an investigational agent within 28 days of first dosing with study treatment.
4. Subject is pregnant or breastfeeding.
5. Subject has active cerebrospinal fluid (CSF) involvement that requires ongoing intrathecal chemotherapy
6. Previous exposure to a Bruton Tyrosine Kinase (BTK) inhibitor.
7. Subjects with severe hepatic insufficiency, as defined by Child-Pugh Score > 6.
8. Subject is receiving prohibited medications or treatments as listed in the protocol that cannot be discontinued/replaced by an alternative therapy.
9. Subject requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists within 14 days of first dose of study drug. Subjects requires or is taking direct oral anticoagulants within 7 days of first dose of study drug.
10. Subject requires treatment with proton pump inhibitors. Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
11. Subject is currently receiving any chemotherapy, anticancer immunotherapy.
12. Subject has clinically significant cardiovascular disease such as ventricular dysfunction, symptomatic coronary artery disease, uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association (NYHA) Functional Classification at screening. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.
13. Subject has familial short QT syndrome.
14. Subject has a history of malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass that is likely to affect absorption.
15. Subject has a known history of infection with HIV or any uncontrolled active significant infection.
16. Subject has a known history of drug-specific hypersensitivity or anaphylaxis to acalabrutinib (including active ingredient or excipient components).
17. Subject has active bleeding or history of bleeding diathesis.
18. Subject has a history of uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP).
19. Subject has a history of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of acalabrutinib.
20. Subject had major surgical procedure within 28 days of first dose of acalabrutinib.
21. Subject who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative PCR result before randomization and must be willing to undergo DNA PCR testing during the study. Subjects who are core antibody positive and viral load negative must receive entecavir Those who are HbsAg-positive, or hepatitis B PCR positive will be excluded.
22. Subjects who are hepatitis C antibody positive must have a negative polymerase chain reaction (PCR) result. Those who are hepatitis C PCR positive will be excluded.
23. Subjects with evidence of disease that investigator decides that is not suitable to enroll in the study.
24. History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML).
25. Received a live virus vaccination within 28 days of first dose of study drug.
26. Any active significant infection.
27. Concurrent participation in another therapeutic clinical trial.
28. Current life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety or put the study at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2030-03-14 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 2 months
  The overall response rate (ORR) will be assessed based on the International Primary CNS Lymphoma Collaborative Group Response assessment criteria. Responder = Partial Response + Complete Response).
  Complete response (CR) as complete disappearance of contrast enhancement on magnetic resonance imaging (MRI), no evidence of ocular lymphoma, negative cerebrospinal fluid (CSF) cytology, and discontinuation of corticosteroid use for at least 2 weeks prior to the evaluation of response. Unconfirmed CR (Cru) is used to characterize radiographic findings that fulfill the criteria for a CR, but the patient remains on corticosteroids, or MRI that continues to show small but persistent enhancing abnormalities possibly related to biopsy or surgery. Partial response (PR) is defined as a 50% decrease in enhancing tumor or residual disease on eye examinations, or persistent or suspicious CSF cytology.

SECONDARY OUTCOMES:
Number of different types of toxicities | 3 years
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).
Progression-free survival (PFS) | 5 years
  Progression-free survival (PFS) is defined from the date of initiating study treatment to the date of disease progression per the International Primary CNS Lymphoma Collaborative Group response assessment criteria or death as a result of any cause.
Complete response (CR) rate | 2 years
  Complete Response (CR) is defined using the International Primary CNS Lymphoma Collaborative Group response assessment criteria for primary CNS lymphoma.
Duration of response (DoR) | 2 years
  Duration of response (DoR) is defined as time from documentation of tumor response to disease progression according to the International Primary CNS Lymphoma Collaborative Group response assessment criteria.
Overall Survival (OS) | 5 years
  OS will be measured from the date of initiating study treatment to the date of death or 5 years (whichever is first). Subjects who have not died by the analysis data cut-off date will be censored at their last date of contact.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dittus, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Moffit Cancer Center, Tampa, Florida
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University,The Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

REFERENCES:
- See also: University of North Carolina - Lineberger Comprehensive Cancer Center - Clinical Trials — https://unclineberger.org/research/